CLINICAL TRIAL: NCT06827392
Title: Evaluation of the Protective Effect of Three Laboratoire VICHY Formulations on the Pigmentation Induced by Visible Light in Comparison with a Non-treated Control Zone
Brief Title: Photoprotection Efficiency with Sunscreen Formulas Under Visible Light Exposure.
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: VCA1601
Record Dates: First submitted 2025-01-13; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Efficiency of Agents; Against Pigmentation Induced by Visible Light Exposures
Keywords: Photoprotection; Sunscreen; Visible Light (VL); Pigmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To evaluate the protective effect of three Laboratoire VICHY formulations on the pigmentation caused by visible light in comparison to a non-treated control zone in healthy volunteers

DETAILED DESCRIPTION:
The sunscreens usually used as photoprotectors are known to protect in the UV domain (UVB and UVA). However, until recently visible light (400-700 nm) was considered as devoid of any photobiological effects on cutaneous tissue. Over the last two decades, with the development of photodynamic therapies and various dermatological treatments using visible laser light, several studies have reconsidered the cutaneous effect of visible light on the skin, in particular the induction of pigmentation.

The aim of this study was to assess the ability of sunscreens with a protective efficacy in the UV domain to prevent the pigmentation induced by Visible Light.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject of both sexes, aged from 18 to 50 years, of phototype IIIb, IV or V on the Fitzpatrick scale (1988),
* Subject in good health having a normal results at the physical examination and having medical antecedents compatible with the study requirements,
* Woman of childbearing potential using a reliable means of contraception (contraceptive pill, contraceptive implant, IUD, bilateral tubal ligature/section, condoms) and agreeing to not change her method of contraception from one month before the start of the study and for the entire duration of the study,
* Healthy woman of non-childbearing potential, that is post-menopausal (absence of menstrual bleeding for one year prior to screening, hysterectomy or bilateral ovariectomy),
* Subject having signed and dated the informed consent form before any action connected to the study was performed,
* Subject willing and able to follow all the study procedures and complete the whole study,
* Subject affiliated to a social security system (according to French legislation: Law 2004-806 and its implementing decree n°2006-477 of 26 April 2006).

Exclusion Criteria:

* Woman who was pregnant or lactating or who planned to become pregnant during the study period,
* Subject having an underlying pathology, or a surgical, physical or medical status which, according to the investigator, could interfere with the interpretation of the study results, such as:

  * A history of dermatological problems (e.g. psoriasis, eczema, urticaria..) or a suspicion/history of allergies to cosmetics or adhesives,
  * All systemic or local pathologies,
  * Skin anomalies (e.g. scars, hirsutism, tattoos…) on the test zones test (middle part of the back),
* Subject having been exposed excessively to ultraviolet light (UV) either natural (sun) or artificial (tanning salon) during the 4 weeks before the screening visit or who planned to expose himself/herself during the study,
* Subject having antecedent or current pathologies induced or aggravated by exposure to light or having abnormal reactions to sunlight (e.g. photosensitive dermatitis, polymorphous light eruption, solar urticaria, systemic lupus erythematosus, dermatomyositis),
* Subject having taken a systemic treatment of more than 5 days during the month preceding inclusion (steroids, non-steroidal anti-inflammatories including aspirin, insulin, anti-histamines, anti-hypertensive drugs, antibiotics such as quinolones, tetracyclines, thiazides and fluoroquinolones, and all photosensitising treatments) or any other treatment capable of inducing an abnormal response to UV or visible light (vitamin A derivatives, psoralen, aminolevulinic acid derivatives…) or who planned to take these treatments during the study,
* Subject who had applied a local treatment on the back for more than 2 days during the 2 weeks preceding inclusion (steroids, non-steroidal anti-inflammatories,, anti-histamines, antibiotics) and any cosmetic products in the 24 hours preceding inclusion,
* Subject with clinically significant allergic antecedents, particularly to components of the test products
* Person requiring enhanced protection (person deprived of liberty, minor, placed under guardianship),
* Subject being in a situation which, according to the opinion of the Investigator, would have interfered with an optimal participation in the study
* Subject participating in, or having participated in, another clinical study during the month preceding inclusion,
* Subject unable to communicate effectively with the investigator or not able to follow the study imperatives.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults meeting the inclusion and exclusion criteria and willing to adhere to the protocol and study procedures
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

PRIMARY OUTCOMES:
Biophysical non-invasive assessment of skin color by using Chromameter® between the exposed zone (ZE) and non-exposed zone (ZNE) | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4 and Day 5 (24 hours after each Visible Light exposure).
  Individual Typologic Angle (ITA° - calculated value),

SECONDARY OUTCOMES:
Clinical investigator's assessment by using clinical scale | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4 and Day 5 (24 hours after each Visible Light exposure).
  Visual scoring of pigmentation, using a pigmentation 11-point scale with 0 (No pigmentation), 1 (Doubtful), 2 (Very pale brown -), 3 (Very pale brown), 4 (Very pale brown +), 5 (Pale brown -), 6 (Pale brown), 7 (Pale brown +), 8 (Brown -), 9 (Brown), 10 (Brown +) Visual scoring of erythema, using an erythema 4-point scale with 0 (Absent), 0.5 (Doubtful), 1 (Weak but well-defined erythema), 2 (Moderate), 3 (Severe)
Safety / Local tolerance | From the informed consent signature date until the end of the study (Day 5)
  Safety was assessed by recording Adverse Events, including cutaneous reactions (local intolerance)
Biophysical non-invasive assessment of skin color by using Chromameter® between the exposed zone (ZE) and non-exposed zone (ZNE) | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4 and Day 5 (24 hours after each Visible Light exposure).
  Pigmentation (Delta E, Delta L* and Delta b* - calculated values)
Biophysical non-invasive assessment of skin color by using Chromameter® between the exposed zone (ZE) and non-exposed zone (ZNE) | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4 and Day 5 (24 hours after each Visible Light exposure).
  Erythema (Delta a* - calculated value).

CONTACTS AND LOCATIONS:
Locations (1):
- CPCAD (Centre de Pharmacologie Clinique Appliquée à la Dermatologie), Nice, France

IPD SHARING:
Plan to Share IPD: No